CLINICAL TRIAL: NCT04723030
Title: Carrilizumab Combined With Apatinib Mesylate and Radiotherapy and Chemotherapy for the Transformation of Locally Advanced Pancreatic Cancer.
Brief Title: The Transformation of Locally Advanced Pancreatic Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, vice president, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BJ-BC-PanC-II-003
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: Carrilizumab；Apatinib mesylate；Locally progressive pancreatic cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- carleilizumab in combination with apathy mesylate and chemoradiotherapy (paclitaxel (albumin-bound) (Experimental): Carilizumab was administered every 2 weeks. The patients were orally taken apatinib after meals and evaluated by DLT(3+3) in the first 2 cycles.The drugs were stopped for 2 weeks after the start of radiotherapy.Before radiotherapy, patients received 2 cycles of karyolizumab combined with apartinib and chemotherapy. Radiotherapy was performed in the first week of cycle 3 with a total dose of 30Gy in five doses within one week.Imaging evaluation was conducted once every 6 weeks. If the patients met the indications for surgical resection, the treatment was stopped.
  Interventions: Drug: carleilizumab+apathy mesylate+radiotherapy+paclitaxel (albumin-bound)

INTERVENTIONS:
Drug: carleilizumab+apathy mesylate+radiotherapy+paclitaxel (albumin-bound) — Carrilizumab ：200mg,q2w; Apatinib :250mg,d1; which is taken continuously for 5 days and stopped for 2 days, and stopped for 2 weeks after radiotherapy.
  Taxol :125mg/m2,q2w; Gemcitabine :1000mg/m2, q2w; cisplatin :25mg/m2, q2w; Radiotherapy:30Gy, divided into five times and completed within one week.

SUMMARY:
This trial will explore the efficacy and safety of camrelizumab combined with apatinib mesylate and radiotherapy and chemotherapy (paclitaxel (albumin binding) combined with gemcitabine and cisplatin) in the treatment of locally advanced pancreatic cancer in patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
This trial is a prospective, observational, single-center, single-arm clinical research.Conversion treatment lasted for a total of 12 weeks, with one treatment cycle every two weeks.Carilizumab was administered every 2 weeks.

The patients were orally taken apatinib after meals and evaluated by DLT(3+3) in the first 2 cycles.The drugs were stopped for 2 weeks after the start of radiotherapy.Before radiotherapy, patients received 2 cycles of karyolizumab combined with apartinib and chemotherapy. Radiotherapy was performed in the first week of cycle 3 with a total dose of 30Gy in five doses within one week.Imaging evaluation was conducted once every 6 weeks. If the patients met the indications for surgical resection, the treatment was stopped

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, both male and female;
2. According to the clinical symptoms, imaging examination, tumor markers and other auxiliary examinations or biopsy results, it was diagnosed as locally progressive pancreatic ductal adenocarcinoma.
3. According to NCCN 2020 V1, locally advanced pancreatic cancer is defined as: 1) no distant metastasis; 2) Arteries: pancreatic head/uncinate process: solid tumors contact superior mesenteric artery > 180; Solid tumors contact abdominal trunk > 180; Solid tumor contacts the first jejunum branch of superior mesenteric artery. Pancreatic body and tail: solid tumors contact superior mesenteric artery or abdominal trunk > 180; Solid tumor touches abdominal trunk and invades aorta. Vein: The superior mesenteric vein/portal vein cannot be reconstructed due to tumor invasion or occlusion (possibly due to tumor or non-tumor embolus).
4. According to the evaluation standard of solid tumor remission (RECIST1.1), there is at least one measurable lesion in imaging diagnosis;
5. Never received local or systemic anti-tumor treatment before, including surgery, chemotherapy, radiotherapy, immunization and targeted therapy;
6. ECOG score is 0 ~ 1;
7. Conscious, can cooperate with positioning, positioning, treatment and respiratory motion control;
8. The main organs function normally, and there are no serious blood, heart, lung, liver, kidney, bone marrow and other abnormal functions and immunodeficiency diseases. Laboratory examination meets the following requirements (no blood components or cell growth factor drugs are allowed to be used within 14 days before the first medication):

   A. hemoglobin ≥ 90g/l; B. absolute neutrophil count ≥ 1.5× 109/l; C. platelet count ≥ 100× 109/l; D. Serum albumin ≥ 28 g/L D. Total bilirubin ≤ 1.5 times the upper limit of normal value; E.ALT and AST ≤ 2.5 times the upper limit of normal value; F. AKP ≤ 2.5 times the normal value; G. serum creatinine ≤ 1 times the upper limit of normal value; H. thyroid stimulating hormone (TSH)≤ 1 times the normal value (if abnormal, FT3 and FT4 levels should be investigated at the same time; if FT3 and FT4 levels are normal, they can be enrolled in the group).
9. Non-surgical sterilization or women of childbearing age need to adopt a medically approved contraceptive measure (such as intrauterine device, contraceptive pill or condom) during the research treatment period and within 3 months after the end of the research treatment period, and the patient voluntarily participates and signs the informed consent form;
10. It is expected that the compliance is good, and the curative effect and adverse reactions can be followed up according to the requirements of the plan.

Exclusion Criteria:

1. Patients with pancreatic cancer who invaded adjacent organs or distant metastasis were found by imaging examination;
2. The patient has any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; Patients with vitiligo; Asthma has been completely relieved in childhood and can be included without any intervention after adults; Asthma in which patients need bronchodilators for medical intervention cannot be included);
3. The patient is using immunosuppressant or systemic hormone therapy to achieve immunosuppression (dose > 10mg/ day prednisone or other therapeutic hormones), and continues to use it within 2 weeks before entering the group;
4. It is known that there is a history of central nervous system metastasis or hepatic encephalopathy;
5. Suffering from hypertension, and can not be well controlled by antihypertensive drug treatment (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg);
6. There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) heart failure above 1)NYHA2 grade 2; (2) unstable angina pectoris; (3) myocardial infarction occurred within one year; (4) clinically significant supraventricular or ventricular arrhythmia needs treatment or intervention; (5)QTc>450ms (male); QTc>470ms (female);
7. Abnormal coagulation function (INR>2.0, PT>16s), bleeding tendency or receiving thrombolytic or anticoagulant therapy, allowing preventive use of low-dose aspirin and low-molecular-weight heparin;
8. In the first 3 months of randomization, there have been bleeding symptoms with significant clinical significance or clear bleeding tendency, such as daily cough/hemoptysis of 2.5ml or more, gastrointestinal bleeding, esophageal varices with bleeding risk, hemorrhagic gastric ulcer or vasculitis, etc. If stool occult blood is positive in baseline period, it can be re-examined. If it is still positive after re-examination, gastroscopy is needed. If gastroscopy indicates severe esophageal varices, it cannot be enrolled in the group (3 months before enrollment.
9. Arterial/venous thrombosis events occurring within the first 6 months, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism, etc.;
10. Known hereditary or acquired bleeding and thrombotic tendencies (such as blood friend patients, coagulation dysfunction, thrombocytopenia, etc.);
11. Urine routine prompts urine protein ≥++and it is confirmed that the amount of urine protein in 24 hours is > 1.0 g;
12. patients with active infection, fever of unknown origin ≥38.5℃ within 7 days before medication, or white blood cell count > 15× 109/l at baseline; 13 patients with congenital or acquired immunodeficiency (such as HIV infection);

14.HBV DNA>2000 IU/ml (or 104 copies/ml); Or HCV RNA>103 copies/ml; Or HBsAg+ and anti-HCV antibody positive patients; 15. The patient has suffered from other malignant tumors in the past 3 years or at the same time (except the cured skin basal cell carcinoma and cervical carcinoma in situ); 16. Vaccination of live vaccine within less than 4 weeks before the study medication or during the study period; 17. There are peripheral neuropathy of grade > 1; 18. Can not cooperate with positioning, positioning, treatment and respiratory motion control; 19. Suffering from uncontrollable mental illness; 20. It is known that there is a history of psychotropic drug abuse or drug abuse; According to the researcher's judgment, the patient has other factors that may affect the research results or lead to the forced termination of the research, such as alcoholism, drug abuse, other serious diseases (including mental diseases) that need to be treated together, serious laboratory examination abnormalities, family or social factors, etc., which will affect the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate(ORR) | 2 years
  The proportion of patients whose tumor volume has reduced to a predetermined value and can maintain the minimum time limit.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 2 years
  The date of first treatment until the date of progression using the RECIST 1.1 criteria, or death due to any cause, whichever comes first.
Descending success rate | Up to 2 years
  Number of patients meeting the resectability criteria of NCCN 2020 V1
R0 resection rate | Up to 2 years
  Number of patients meeting the R0 resection standard.
R1 resection rate | Up to 2 years
  Number of patients meeting the R1 resection standard.
Subject safety | Up to 2 years
  Number of Adverse Events using NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: LIN SHEN, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality
  - Peking University Cancer Hospital & Institute, Beijing